CLINICAL TRIAL: NCT00159211
Title: Evolution of Abdominal Adipose Tissue Distribution in Type 2 Diabetic Patients Treated During 6 Months With Pioglitazone or Insulin, in Association With Metformin or Sulfonylurea.
Brief Title: Abdominal Adipose Tissue Distribution in Type 2 Diabetic Patients Treated During 6 Months With Pioglitazone or Insulin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion was finished
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Laboratoires Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P031006
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2007-11-08 (Estimated); Status verified 2007-04

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): UMULINE NPH at bed time
  Interventions: Drug: UMULINE NPH
- 2 (Experimental): pioglitazone 30 mg
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: UMULINE NPH — UMULINE NPH at bed time with a increasing dose up to get a fasting glycemia under 1.1 g/l
  Arms: 1
Drug: pioglitazone — 30mg daily. After 2 months, if HbA1c has not decreased at least of 1%, the dosage should be increased to 45 mg daily
  Arms: 2

SUMMARY:
In type 2 diabetic patients with poor glycemic control despite maximum "classic" oral treatment, bed time insulin therapy may lead to a parallel increase in abdominal visceral and subcutaneous fat, whereas pioglitazone treatment should lead to a stability (or even a decrease ) in visceral and an increase in subcutaneous abdominal fat. As visceral fat mass is correlated with insulin-resistance and cardio-vascular risk, the evolution of visceral abdominal fat in type 2 diabetic patients is of great importance.

Main objective:

To compare visceral and subcutaneous abdominal fat compartment after a six-month bed time insulin or pioglitazone treatment in type 2 diabetic patients with poor glycemic control despite a maximal oral treatment with metformin and sulfonylureas.

The study hypothesis is that quantity of visceral and subcutaneous abdominal adipose tissue should differently evolute comparing a 6 month treatment with pioglitazone® (30 or 45mg/j) or NPH " bed-time " insulin (0.2u/kg/

DETAILED DESCRIPTION:
In type 2 diabetic patients with poor glycemic control despite maximum "classic" oral treatment, bed time insulin therapy may lead to a parallel increase in abdominal visceral and subcutaneous fat, whereas pioglitazone treatment should lead to a stability (or even a decrease ) in visceral and an increase in subcutaneous abdominal fat. As visceral fat mass is correlated with insulin-resistance and cardio-vascular risk, the evolution of visceral abdominal fat in type 2 diabetic patients is of great importance.

The study hypothesis is that quantity of visceral and subcutaneous abdominal adipose tissue should differently evolute comparing a 6 month treatment with pioglitazone® (30 or 45mg/j) or NPH " bed-time " insulin (0.2u/kg/

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* BMI= 26kg/m2
* Maximal treatment with metformin and sulfonylurea
* HbA1c between 7.5 and 9.5%

Exclusion Criteria:

* Anterior treatment with glitazones
* Anterior treatment with insulin
* Known heart failure
* Hepatopathy
* Renal filtration less than 60ml/min, Hb<10g/dl
* Corticoids treatment

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-05; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Abdominal adipose tissue (on scan) variation at 6 month | 6 months

SECONDARY OUTCOMES:
Cellularity of subcutaneous adipose variation tissue at 6 month | 6 months
HbA1c, lipid level, adiponectin, CRP variation at 6 month | 6 months
inflammation gene expression in sub-cutaneous fat | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Agnès Hartemann-Heurtier, MDPHD, Principal Investigator — Assistance Publique des Hôpitaux de Paris Hôpital Pitié Salpêtrière France
Locations (1):
- Sce de Diabétologie, hôpital de la Pitié-salpêtrière, 83bld de l'hôpital, Paris, France

REFERENCES:
- [Derived] Hartemann-Heurtier A, Halbron M, Golmard JL, Jacqueminet S, Bastard JP, Rouault C, Ayed A, Pieroni L, Clement K, Grimaldi A. Effects of bed-time insulin versus pioglitazone on abdominal fat accumulation, inflammation and gene expression in adipose tissue in patients with type 2 diabetes. Diabetes Res Clin Pract. 2009 Oct;86(1):37-43. doi: 10.1016/j.diabres.2009.06.028. Epub 2009 Aug 15. PMID 19683825